CLINICAL TRIAL: NCT05205174
Title: Depth Electrode Detection of Cortical Spreading Depolarization After Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-FY2021-251
Record Dates: First submitted 2021-12-14; First posted 2022-01-25 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Feasibility (Other): This is a preliminary, prospective interventional study to investigate the feasibility of using depth electrodes in conjunction with novel analytical algorithms to detect CSDs in TBI patients.
  Interventions: Device: depth electrodes

INTERVENTIONS:
Device: depth electrodes — The study will be conducted at a single center, in TBI patients requiring neurosurgical intervention in the form of EVD placement. During neurosurgical intervention at the bedside in the Intensive Care Unit (ICU), a single depth electrode will be placed in the brain adjacent to the EVD catheter in the same burr hole. After EVD and depth electrode placement, continuous recording of ECoG activity as well as relevant physiological parameters will be performed for the duration of clinically indicated invasive neuromonitoring in accordance with the standard of care for TBI patients. A single recording station is currently available for data collection, therefore, with an anticipated average recording period of 14 days, the study will take greater than 210 days to complete for a total of 15 patients.

SUMMARY:
Preliminary evaluation of depth electrode recording and novel algorithms to determine Cortical Spreading Depolarization's (CSD) following traumatic brain injury (TBI) requiring neurosurgical intervention.

DETAILED DESCRIPTION:
During the standard of care External Ventricular Drain (EVD) placement, a depth electrode with minimal modification to the standard surgical procedure will be placed. This will allow electrocorticogram (ECoG) recordings. An ECoG will be reviewed by a study Neurosurgeon to understand the association between cortical spreading depression and pathological findings on imaging. The recordings help create a novel algorithm in order to detect CSD's. This may ultimately provide significant benefit to society through the diagnosis and treatment of secondary injury associated with traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Patient recommended to undergo EVD placement for the monitoring and possible treatment of Intracranial pressure (ICP) after TBI

Exclusion Criteria:

* Contaminated scalp lacerations
* Known systemic infection
* Non-English speaking
* Fixed, uncorrectable coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-12-03 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Detecting CSDs in TBI patients | 2 years
  The primary endpoint is to determine the feasibility of using depth electrodes in conjunction with novel analytical algorithms to detect CSDs in TBI patients. A single depth electrode will be placed at the same time the EVD is performed. ECoG recordings from each patient will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, MD, Principal Investigator — University of Minnesota
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No